CLINICAL TRIAL: NCT06906731
Title: An Open-label, Multicenter Phase I/II Study of Safety, Tolerability,Pharmacokinetics and Efficacy of SHR-9803 for Injection in Patients With Advanced Solid Tumors
Brief Title: A Study of SHR-9803 for Injection in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-9803-101
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-9803 (Experimental): SHR-9803
  Interventions: Drug: SHR-9803

INTERVENTIONS:
Drug: SHR-9803 — SHR-9803

SUMMARY:
This is an open label, multi-center, multiple doses Phase I/II study to evaluate the safety, tolerability ,pharmacokinetics and efficacy of SHR-9803 for injection in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent.
2. 18-75 years old, no gender limitation.
3. Eastern Cooperative Oncology Group (ECOG) score: 0-1
4. With a life expectancy ≥ 3 months.
5. Pathologically diagnosed advanced solid tumor.
6. At least one measurable lesion according to RECIST v1.1.
7. Adequate bone marrow reserve and organ function.
8. Contraception is required during clinical trials, and pregnancy tests must be negative for women of childbearing age within 7 days before the first dose.

Exclusion Criteria:

1. Have untreated central nervous system metastasis; or have meningeal metastasis or spinal cord compression;
2. Uncontrolled clinically symptomatic pleural effusion, pericardial effusion, or ascites;
3. Previous or co-existing malignancies；
4. Severe bone damage caused by bone metastasis， including uncontrolled tumor-related pain;
5. Have active or prior documented autoimmune disease;
6. Have used corticosteroids (> 10 mg/day of prednisone or equivalent) or other immunosuppressive agents for systemic treatment within 2 weeks;
7. With poorly controlled or severe cardiovascular disease;
8. A history of interstitial pneumonia/non-infectious pneumonia;
9. Severe infection 1 month before the first dose;
10. Active hepatitis B or hepatitis C, or with a history of immunodeficiency;
11. With a history of inflammatory bowel disease, or those who have experienced intestinal obstruction or gastrointestinal perforation within 3 months prior to the first dose;
12. Have received more than 30 Gy of pulmonary radiation therapy within 6 months prior to the first dose; Have received major surgery，Systemic chemotherapy, endocrine therapy, monoclonal antibody therapy, macromolecular targeted therapy or other investigational products within 4 weeks; or palliative radiotherapy within 2 weeks; or oral small-molecule targeted drugs within five half-lives;
13. Have not recovered from the toxicities and/or complications of previous interventions to NCI-CTCAE Grade ≤ 1;
14. Received live-attenuated vaccines within 4 weeks prior to the first dose.
15. Known to have had an allergic reaction to other monoclonal antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity（Ia） | Screening up to the end of phase Ia, an average of 6 months
Dose Limited Toxicity (Ib) | Screening up to the end of phase Ib, an average of 1 year
Recommended phase II dose(Ib) | Screening up to the end of phase Ib, an average of 2 years
objective response rate(II) | Screening up to study completion, an average of 3 year

SECONDARY OUTCOMES:
Adverse Events, | Screening up to study completion, an average of 3 year;
Disease Control Rate (DCR), | Screening up to study completion, an average of 3 year
Progression-Free Survival (PFS), | Screening up to study completion, an average of 3 year;
Plasma concentration of SHR-9803 | Screening up to study completion, an average of 3 year;

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University cancer hospital, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided